CLINICAL TRIAL: NCT01425814
Title: A Phase IIa, Randomised, Single Dose, Double-blind, Double-dummy, 6 Way Complete Cross-over, Placebo Controlled Clinical Trial to Assess the Efficacy, Safety and Tolerability of 4 Strengths of LAS100977 QD Compared to Placebo and an Active Comparator in Patients With Stable Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Single Dose Study to Assess Efficacy and Safety of 4 Doses of LAS100977 in Chronic Obstructive Pulmonary Disease (COPD) Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M/100977/25; LBC25
Record Dates: First submitted 2011-08-29; First posted 2011-08-30 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm #2 (Experimental): Single dose, double blind treatment period
  Interventions: Drug: LAS100977
- Arm #3 (Experimental): Single dose, double blind treatment period
  Interventions: Drug: LAS100977
- Arm #4 (Experimental): Single dose, double blind treatment period
  Interventions: Drug: LAS100977
- Arm #5 (Active Comparator): Single dose, double blind treatment period
  Interventions: Drug: Reference
- Arm #6 (Placebo Comparator): Single dose, double blind treatment period
  Interventions: Drug: Placebo
- Arm #1 (Experimental): Single dose, double blind treatment period
  Interventions: Drug: LAS100977

INTERVENTIONS:
Drug: LAS100977 — Dry powder inhalation,Once daily, single dose
  Arms: Arm #1
Drug: LAS100977 — Dry powder inhalation,Once daily, single dose
  Arms: Arm #2
Drug: LAS100977 — Dry powder inhalation,Once daily, single dose
  Arms: Arm #3
Drug: LAS100977 — Dry powder inhalation,Once daily, single dose
  Arms: Arm #4
Drug: Reference — Dry powder inhalation (capsule),single dose
  Arms: Arm #5
Drug: Placebo — Dry powder inhalation or Dry powder inhalation (capsule),Once daily, single dose
  Arms: Arm #6

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamics (bronchodilation) of single doses of inhaled LAS100977 in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females aged 40 or older.
2. Patients with a clinical diagnosis of COPD, according to the GOLD guidelines and stable airway obstruction.
3. Patients with a post-salbutamol FEV1 equal to or greater than 30% of the predicted value and less than 80% of the predicted value
4. Post-salbutamol FEV1/FVC < 70% at screening visit.
5. Pre-dose FEV1 value of first treatment period within the range of 80-120% of the FEV1 measured at screening prior to salbutamol inhalation.
6. Current, or ex-cigarette smokers (former) with a smoking history of at least 10 pack-years.
7. Patients whose COPD symptoms at the time of randomisation are stable compared to the Screening visit, according to the investigator's medical judgment.

Exclusion Criteria:

1. History or current diagnosis of asthma.
2. A respiratory tract infection or COPD exacerbation in the six weeks prior to the screening visit.
3. Patients who have been hospitalised for an acute COPD exacerbation in the 3 months prior to screening visit.
4. Clinically significant respiratory conditions other than COPD condition.
5. Clinically significant cardiovascular conditions.
6. Patients unable to properly use a dry powder or pMDI inhaler device or unable to perform acceptable spirometry.
7. Clinically relevant abnormalities laboratory, ECG parameters or physical examination results at the screening evaluation that in the investigator's opinion, preclude study participation.
8. Patients who intend to use any concomitant medication not permitted by this protocol or who have not undergone the required washout period for a particular prohibited medication.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Astbury, PhD, Study Director — AstraZeneca
Locations (8):
- Germany (8):
  - Almirall Investigational Sites#5, Berlin
  - Almirall Investigational Sites#2, Berlin
  - Almirall Investigational Sites#6, Frankfurt
  - Almirall Investigational Sites#3, Großhansdorf
  - Almirall Investigational Sites#7, Hamburg
  - Almirall Investigational Sites#8, Lübeck
  - Almirall Investigational Sites#1, Mainz
  - Almirall Investigational Sites#4, Wiesbaden

REFERENCES:
- [Derived] Beier J, Pujol H, Seoane B, Jimenez E, Astbury C, Massana E, Ruiz S, de Miquel G. Abediterol, a novel long-acting beta2-agonist: bronchodilation, safety, tolerability and pharmacokinetic results from a single-dose, dose-ranging, active-comparator study in patients with COPD. BMC Pulm Med. 2016 Jul 20;16(1):102. doi: 10.1186/s12890-016-0266-5. PMID 27439370
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3969&filename=M-100977-25_CSRsynopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 9 sites in Germany, 8 of which randomized patients
Pre-assignment Details: Screening took place 14±2 days before randomization. After screening, eligible patients entered a run-in period to assess clinical stability. A total of 87 patients were screened, of whom 70 patients were assessed as eligible and randomized; 17 were not randomized due to screening failure (primarily non-fulfillment of inclusion/exclusion criteria)
Groups:
- Sequence A: Indacaterol 150 μg - LAS100977 10 μg - Placebo - LAS100977 0.625 μg - LAS100977 5 μg- LAS100977 2.5 μg
- Sequence B: LAS100977 10 μg - LAS100977 0.625 μg - Indacaterol 150 μg - LAS100977 2.5 μg - Placebo - LAS100977 5 μg
- Sequence C: LAS100977 0.625 μg - LAS100977 2.5 μg - LAS100977 10 μg - LAS100977 5 μg - Indacaterol 150 μg - Placebo
- Sequence D: LAS100977 2.5 μg - LAS100977 5 μg - LAS100977 0.625 μg - Placebo - LAS100977 10 μg - Indacaterol 150 μg
- Sequence E: LAS100977 5 μg - Placebo - LAS100977 2.5 μg - Indacaterol 150 μg - LAS100977 0.625 μg - LAS100977 10 μg
- Sequence F: Placebo - Indacaterol 150 μg - LAS100977 5 μg - LAS100977 10 μg - LAS100977 2.5 μg - LAS100977 0.625 μg
Period: Period 1
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 12 | 11 | 12 | 10 | 12 | 13
Completed | 12 | 10 | 12 | 10 | 12 | 13
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Stability criteria not fulfilled | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 12 | 10 | 12 | 10 | 12 | 13
Completed | 12 | 9 | 12 | 10 | 12 | 13
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Stability criteria not fulfilled | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 12 | 9 | 12 | 10 | 12 | 13
Completed | 12 | 9 | 12 | 10 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 4
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 12 | 9 | 12 | 10 | 12 | 12
Completed | 11 | 9 | 11 | 10 | 12 | 12
Not Completed | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 11 | 9 | 11 | 10 | 12 | 12
Completed | 11 | 9 | 10 | 10 | 12 | 11
Not Completed | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Stability criteria not fulfilled | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Population: All patients who were randomized and received at least one dose of investigational medicinal product
Arm/Group | Overall Population
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1)
Description: Baseline was the average of the two values measured just prior to the administration of the dose of investigational medicinal product at Day 1 of each visit (time points -45 min and -15 min) Trough at Day 2 was computed as the average of the two values measured at 23 and 24 hours after administration of the morning dose of investigational medicinal product on Day 1 At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 and FVC were selected
Time Frame: Day 2
Population: ITT population defined as patients who took at least one dose of investigational medicinal product and had at least a baseline and one post-dose value of FEV1 from at least one treatment period
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Placebo: Single dose administered by inhalation from the Genuair® device and the Breezhaler® inhaler
- LAS100977 0.625 μg; LAS100977 2.5 μg; LAS100977 5 μg; LAS100977 10 μg: Single dose administered by inhalation from the Genuair® device
- Indacaterol 150 μg: Single dose administered by inhalation from the Breezhaler® inhaler
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters | -0.035 (0.024) | 0.066 (0.024) | 0.168 (0.024) | 0.198 (0.024) | 0.223 (0.024) | 0.076 (0.024)
Statistical Analysis 1: Comparison: Placebo vs LAS100977 10 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = 0.259, 95% CI 2-sided [0.219 to 0.298], Standard Error of Mean 0.020
Statistical Analysis 2: Comparison: Placebo vs LAS100977 5 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = 0.233, 95% CI 2-sided [0.194 to 0.273], Standard Error of Mean 0.020
Statistical Analysis 3: Comparison: Placebo vs LAS100977 2.5 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = 0.203, 95% CI 2-sided [0.164 to 0.242], Standard Error of Mean 0.020
Statistical Analysis 4: Comparison: Placebo vs LAS100977 0.625 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = 0.102, 95% CI 2-sided [0.062 to 0.141], Standard Error of Mean 0.020

2. Secondary Outcome: Change From Baseline in Normalised Forced Expiratory Volume in One Second (FEV1) Area Under the Curve
Description: Baseline was the average of the two values measured just prior to the administration of the dose of investigational medicinal product at Day 1 of each visit (time points -45 min and -15 min) At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 and FVC were selected
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters
  Change from baseline in FEV1 AUC0-12 | -0.003 (0.012) | 0.168 (0.021) | 0.243 (0.021) | 0.247 (0.021) | 0.288 (0.022) | 0.134 (0.017)
  Change from baseline in FEV1 AUC0-24 | -0.032 (0.013) | 0.121 (0.021) | 0.205 (0.022) | 0.222 (0.021) | 0.262 (0.024) | 0.104 (0.018)
  Change from baseline in FEV1 AUC12-24 | -0.062 (0.016) | 0.077 (0.023) | 0.166 (0.024) | 0.196 (0.021) | 0.235 (0.021) | 0.073 (0.021)

3. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1)
Description: as for outcome 2
Time Frame: Up to Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters
  Baseline | 1.475 (0.059) | 1.506 (0.065) | 1.472 (0.062) | 1.483 (0.063) | 1.493 (0.065) | 1.488 (0.064)
  Day 1 0.08 hr | -0.005 (0.013) | 0.044 (0.011) | 0.090 (0.011) | 0.085 (0.012) | 0.117 (0.016) | 0.103 (0.014)
  Day 1 0.25 hr | 0.006 (0.013) | 0.087 (0.016) | 0.155 (0.015) | 0.161 (0.015) | 0.191 (0.019) | 0.132 (0.016)
  Day 1 0.5 hr | 0.018 (0.015) | 0.126 (0.019) | 0.186 (0.018) | 0.202 (0.019) | 0.217 (0.021) | 0.150 (0.017)
  Day 1 1 hr | 0.010 (0.015) | 0.151 (0.020) | 0.217 (0.021) | 0.218 (0.018) | 0.240 (0.023) | 0.156 (0.016)
  Day 1 2 hr | 0.002 (0.016) | 0.166 (0.022) | 0.230 (0.021) | 0.245 (0.019) | 0.261 (0.024) | 0.161 (0.019)
  Day 1 3 hr | 0.018 (0.014) | 0.201 (0.022) | 0.287 (0.022) | 0.274 (0.024) | 0.321 (0.023) | 0.184 (0.020)
  Day 1 4 hr | 0.015 (0.014) | 0.225 (0.021) | 0.308 (0.023) | 0.308 (0.024) | 0.341 (0.173) | 0.179 (0.018)
  Day 1 6 hr | -0.005 (0.017) | 0.216 (0.028) | 0.276 (0.024) | 0.276 (0.022) | 0.311 (0.031) | 0.135 (0.018)
  Day 1 8 hr | 0.007 (0.016) | 0.169 (0.025) | 0.260 (0.025) | 0.263 (0.024) | 0.313 (0.025) | 0.124 (0.021)
  Day 1 12 hr | -0.047 (0.017) | 0.115 (0.025) | 0.189 (0.027) | 0.202 (0.027) | 0.271 (0.026) | 0.085 (0.023)
  Day 1 14 hr | -0.067 (0.020) | 0.099 (0.026) | 0.180 (0.026) | 0.214 (0.24) | 0.250 (0.026) | 0.087 (0.022)
  Day 2 23 hr | -0.066 (0.017) | 0.036 (0.023) | 0.134 (0.026) | 0.166 (0.022) | 0.211 (0.030) | 0.050 (0.022)
  Day 2 24 hr | -0.018 (0.019) | 0.093 (0.023) | 0.184 (0.025) | 0.205 (0.021) | 0.236 (0.027) | 0.088 (0.020)
  Day 2 36 hr | -0.020 (0.020) | 0.040 (0.024) | 0.104 (0.022) | 0.083 (0.023) | 0.116 (0.024) | 0.036 (0.021)

4. Secondary Outcome: Absolute Forced Expiratory Volume in One Second (FEV1) Values
Description: At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 and FVC were selected
Time Frame: Up to Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters
  Baseline | 1.475 (0.059) | 1.506 (0.065) | 1.472 (0.062) | 1.483 (0.063) | 1.493 (0.065) | 1.488 (0.064)
  Day 1 0.08 hr | 1.474 (0.060) | 1.549 (0.064) | 1.561 (0.064) | 1.568 (0.062) | 1.610 (0.065) | 1.585 (0.064)
  Day 1 0.25 hr | 1.482 (0.059) | 1.592 (0.064) | 1.627 (0.063) | 1.644 (0.064) | 1.673 (0.066) | 1.620 (0.063)
  Day 1 0.5 hr | 1.494 (0.060) | 1.640 (0.064) | 1.658 (0.063) | 1.685 (0.065) | 1.708 (0.067) | 1.683 (0.065)
  Day 1 1 hr | 1.485 (0.061) | 1.657 (0.066) | 1.688 (0.065) | 1.701 (0.067) | 1.733 (0.069) | 1.624 (0.061)
  Day 1 2 hr | 1.477 (0.061) | 1.671 (0.067) | 1.701 (0.067) | 1.729 (0.067) | 1.754 (0.068) | 1.642 (0.066)
  Day 1 3 hr | 1.494 (0.061) | 1.707 (0.069) | 1.758 (0.068) | 1.758 (0.069) | 1.814 (0.071) | 1.672 (0.066)
  Day 1 4 hr | 1.491 (0.061) | 1.730 (0.068) | 1.780 (0.068) | 1.790 (0.070) | 1.840 (0.073) | 1.677 (0.067)
  Day 1 6 hr | 1.477 (0.062) | 1.721 (0.070) | 1.748 (0.070) | 1.759 (0.069) | 1.804 (0.074) | 1.623 (0.065)
  Day 1 8 hr | 1.490 (0.062) | 1.674 (0.070) | 1.732 (0.070) | 1.746 (0.070) | 1.806 (0.073) | 1.612 (0.065)
  Day 1 12 hr | 1.428 (0.061) | 1.629 (0.069) | 1.660 (0.066) | 1.686 (0.068) | 1.761 (0.073) | 1.565 (0.067)
  Day 1 14 hr | 1.409 (0.061) | 1.605 (0.068) | 1.646 (0.068) | 1.693 (0.069) | 1.740 (0.072) | 1.585 (0.065)
  Day 2 23 hr | 1.411 (0.061) | 1.542 (0.068) | 1.606 (0.070) | 1.649 (0.070) | 1.701 (0.074) | 1.538 (0.064)
  Day 2 24 hr | 1.464 (0.062) | 1.599 (0.070) | 1.655 (0.071) | 1.688 (0.070) | 1.726 (0.073) | 1.576 (0.066)
  Day 2 36 hr | 1.464 (0.064) | 1.564 (0.068) | 1.575 (0.068) | 1.566 (0.069) | 1.607 (0.069) | 1.524 (0.064)

5. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in One Second (FEV1)
Description: as for outcome 2
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters | 0.098 (0.016) | 0.290 (0.025) | 0.351 (0.022) | 0.350 (0.023) | 0.391 (0.024) | 0.263 (0.019)

6. Secondary Outcome: Time to Peak Forced Expiratory Volume in One Second (FEV1)
Description: as for outcome 4
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Hours | 2.5 (0.2) | 3.4 (0.2) | 3.5 (0.2) | 3.7 (0.2) | 4.0 (0.2) | 2.9 (0.2)

7. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (FVC)
Description: as for outcome 1
Time Frame: Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters | -0.079 (0.044) | 0.067 (0.044) | 0.180 (0.044) | 0.217 (0.044) | 0.254 (0.044) | 0.088 (0.044)

8. Secondary Outcome: Change From Baseline in Normalised Forced Vital Capacity (FVC) Area Under the Curve
Description: as for outcome 2
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters
  Change from baseline in FVC AUC0-12 | 0.026 (0.026) | 0.253 (0.037) | 0.297 (0.036) | 0.306 (0.034) | 0.372 (0.037) | 0.237 (0.033)
  Change from baseline in FVC AUC0-24 | -0.034 (0.027) | 0.170 (0.036) | 0.253 (0.039) | 0.272 (0.035) | 0.328 (0.038) | 0.175 (0.033)
  Change from baseline in FVC AUC12-24 | -0.096 (0.031) | 0.089 (0.039) | 0.208 (0.045) | 0.236 (0.039) | 0.284 (0.042) | 0.114 (0.037)

9. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: as for outcome 2
Time Frame: Up to Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters
  Baseline | 3.165 (0.101) | 3.195 (0.104) | 3.137 (0.102) | 3.153 (0.094) | 3.212 (0.108) | 3.190 (0.106)
  Day 1 0.08 hr | 0.048 (0.026) | 0.098 (0.027) | 0.166 (0.034) | 0.178 (0.027) | 0.267 (0.040) | 0.221 (0.034)
  Day 1 0.25 hr | 0.004 (0.027) | 0.140 (0.033) | 0.193 (0.037) | 0.212 (0.033) | 0.264 (0.036) | 0.192 (0.035)
  Day 1 0.5 hr | 0.127 (0.085) | 0.191 (0.035) | 0.232 (0.037) | 0.263 (0.036) | 0.277 (0.037) | 0.246 (0.036)
  Day 1 1 hr | 0.052 (0.029) | 0.242 (0.041) | 0.263 (0.043) | 0.241 (0.036) | 0.289 (0.042) | 0.246 (0.041)
  Day 1 2 hr | 0.036 (0.035) | 0.224 (0.041) | 0.0269 (0.040) | 0.300 (0.035) | 0.303 (0.042) | 0.244 (0.036)
  Day 1 3 hr | 0.020 (0.026) | 0.248 (0.044) | 0.338 (0.041) | 0.325 (0.041) | 0.392 (0.039) | 0.274 (0.037)
  Day 1 4 hr | 0.016 (0.030) | 0.297 (0.042) | 0.379 (0.039) | 0.337 (0.042) | 0.402 (0.035) | 0.254 (0.035)
  Day 1 6 hr | 0.036 (0.034) | 0.340 (0.048) | 0.327 (0.044) | 0.348 (0.042) | 0.415 (0.044) | 0.231 (0.036)
  Day 1 8 hr | 0.048 (0.037) | 0.263 (0.045) | 0.309 (0.044) | 0.335 (0.040) | 0.425 (0.050) | 0.266 (0.046)
  Day 1 12 hr | -0.035 (0.038) | 0.198 (0.048) | 0.259 (0.046) | 0.272 (0.050) | 0.329 (0.048) | 0.182 (0.047)
  Day 1 14 hr | -0.110 (0.043) | 0.107 (0.047) | 0.236 (0.050) | 0.266 (0.043) | 0.315 (0.046) | 0.148 (0.045)
  Day 2 23 hr | -0.093 (0.037) | 0.039 (0.042) | 0.153 (0.050) | 0.187 (0.044) | 0.244 (0.051) | 0.063 (0.041)
  Day 2 24 hr | -0.076 (0.035) | 0.090 (0.039) | 0.186 (0.038) | 0.207 (0.039) | 0.243 (0.046) | 0.100 (0.040)
  Day 2 36 hr | -0.023 (0.037) | 0.063 (0.040) | 0.114 (0.045) | 0.059 (0.038) | 0.140 (0.040) | 0.084 (0.040)

10. Secondary Outcome: Absolute Forced Vital Capacity (FVC) Values
Description: as for outcome 4
Time Frame: Up to Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters
  Baseline | 3.165 (0.101) | 3.195 (0.104) | 3.137 (0.102) | 3.153 (0.094) | 3.212 (0.108) | 3.190 (0.106)
  Day 1 0.08 hr | 3.205 (0.106) | 3.293 (0.112) | 3.318 (0.105) | 3.331 (0.100) | 3.479 (0.116) | 3.418 (0.117)
  Day 1 0.25 hr | 3.169 (0.098) | 3.335 (0.109) | 3.329 (0.102) | 3.365 (0.100) | 3.455 (0.111) | 3.382 (0.107)
  Day 1 0.5 hr | 3.292 (0.126) | 3.399 (0.110) | 3.368 (0.105) | 3.417 (0.101) | 3.488 (0.112) | 3.441 (0.110)
  Day 1 1 hr | 3.217 (0.104) | 3.436 (0.110) | 3.400 (0.107) | 3.394 (0.102) | 3.501 (0.114) | 3.415 (0.111)
  Day 1 2 hr | 3.201 (0.101) | 3.418 (0.111) | 3.406 (0.107) | 3.454 (0.102) | 3.514 (0.109) | 3.415 (0.108)
  Day 1 3 hr | 3.185 (0.099) | 3.443 (0.109) | 3.475 (0.106) | 3.478 (0.103) | 3.603 (0.116) | 3.464 (0.110)
  Day 1 4 hr | 3.181 (0.101) | 3.492 (0.108) | 3.516 (0.103) | 3.478 (0.099) | 3.608 (0.114) | 3.448 (0.110)
  Day 1 6 hr | 3.220 (0.097) | 3.535 (0.118) | 3.464 (0.109) | 3.501 (0.109) | 3.626 (0.119) | 3.421 (0.109)
  Day 1 8 hr | 3.232 (0.103) | 3.458 (0.114) | 3.445 (0.110) | 3.488 (0.107) | 3.636 (0.122) | 3.469 (0.116)
  Day 1 12 hr | 3.130 (0.105) | 3.406 (0.118) | 3.396 (0.108) | 3.425 (0.105) | 3.534 (0.119) | 3.367 (0.115)
  Day 1 14 hr | 3.055 (0.107) | 3.302 (0.112) | 3.359 (0.111) | 3.411 (0.107) | 3.520 (0.118) | 3.348 (0.118)
  Day 2 23 hr | 3.075 (0.108) | 3.233 (0.111) | 3.290 (0.107) | 3.341 (0.107) | 3.448 (0.117) | 3.257 (0.106)
  Day 2 24 hr | 3.095 (0.103) | 3.284 (0.109) | 3.323 (0.104) | 3.360 (0.102) | 3.447 (0.110) | 3.295 (0.107)
  Day 2 36 hr | 3.145 (0.102) | 3.289 (0.109) | 3.251 (0.108) | 3.212 (0.102) | 3.345 (0.110) | 3.274 (0.105)

11. Secondary Outcome: Change From Baseline in Peak Forced Vital Capacity (FVC)
Description: as for outcome 2
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters | 0.332 (0.050) | 0.484 (0.050) | 0.523 (0.050) | 0.532 (0.050) | 0.575 (0.050) | 0.470 (0.050)

12. Secondary Outcome: Time to Peak Forced Vital Capacity (FVC)
Description: as for outcome 4
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Hours | 2.4 (0.3) | 3.6 (0.3) | 3.4 (0.2) | 3.1 (0.2) | 3.6 (0.3) | 2.6 (0.3)

13. Secondary Outcome: Change From Baseline in Inspiratory Capacity (IC)
Description: Baseline was the average of the two values measured just prior to the administration of the dose of investigational medicinal product at Day 1 of each visit (time points -45 min and -15 min) At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS
Time Frame: Up to Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters
  Baseline | 2.240 (0.082) | 2.239 (0.078) | 2.234 (0.075) | 2.254 (0.077) | 2.237 (0.077) | 2.246 (0.076)
  Day 1 4 hr | 0.004 (0.037) | 0.260 (0.039) | 0.239 (0.040) | 0.316 (0.043) | 0.370 (0.043) | 0.215 (0.036)
  Day 2 24 hr | -0.047 (0.040) | 0.110 (0.037) | 0.157 (0.037) | 0.174 (0.038) | 0.273 (0.046) | 0.136 (0.035)

14. Secondary Outcome: Absolute Inspiratory Capacity (IC) Values
Description: At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS
Time Frame: Up to Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Number analyzed (Participants) | 68 | 67 | 66 | 66 | 67 | 68
Liters
  Baseline | 2.240 (0.082) | 2.239 (0.078) | 2.234 (0.075) | 2.254 (0.077) | 2.237 (0.077) | 2.246 (0.076)
  Day 1 4 hr | 2.279 (0.076) | 2.504 (0.081) | 2.473 (0.083) | 2.548 (0.088) | 2.623 (0.088) | 2.447 (0.079)
  Day 2 24 hr | 2.203 (0.074) | 2.374 (0.082) | 2.398 (0.085) | 2.402 (0.081) | 2.543 (0.086) | 2.380 (0.077)

ADVERSE EVENTS:
Time Frame: Up to 14 (±2) days after the last investigational medicinal product administration
Arm/Group | Placebo | LAS100977 0.625 μg | LAS100977 2.5 μg | LAS100977 5 μg | LAS100977 10 μg | Indacaterol 150 μg
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/67 | 0/66 | 1/66 | 1/67 | 0/68
Other Adverse Events (participants affected / at risk) | 2/68 | 4/67 | 1/66 | 1/66 | 2/67 | 5/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | LAS100977 0.625 μg (N=67) | LAS100977 2.5 μg (N=66) | LAS100977 5 μg (N=66) | LAS100977 10 μg (N=67) | Indacaterol 150 μg (N=68)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | LAS100977 0.625 μg (N=67) | LAS100977 2.5 μg (N=66) | LAS100977 5 μg (N=66) | LAS100977 10 μg (N=67) | Indacaterol 150 μg (N=68)
Nasopharyngitis (Infections and infestations) | 2 | 4 | 1 | 1 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication and/or presentation, whether complete or partial, of any part of the data or results of this trial will be subjected to revision and written agreement between the investigator and Sponsor